CLINICAL TRIAL: NCT00890630
Title: Intracervical Catheters for Induction of Labour in Women With Prelabour Rupture of Membranes at Term: A Pilot Study.
Brief Title: Intracervical Catheters for Induction of Labour in Women With Prelabour Rupture of Membranes at Term
Acronym: IC-PROM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate Patient Recruitment.
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Dr. Amie Cullimore, Faculty of Health Sciences, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-3265
Record Dates: First submitted 2009-04-27; First posted 2009-04-30 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Fetal Membranes, Premature Rupture; Induced Labor
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Active Comparator): Induction of Labour with Oxytocin Alone
  Interventions: Drug: Oxytocin
- Intracervical Catheter (Experimental): Insertion of an Intracervical Balloon Catheter plus administration of oxytocin for labour induction.
  Interventions: Procedure: Intracervical Balloon Catheter; Drug: Oxytocin

INTERVENTIONS:
Procedure: Intracervical Balloon Catheter — Intracervical insertion of an 80cc Double-Balloon Catheter.
  Arms: Intracervical Catheter
Drug: Oxytocin — IV Oxytocin infusion, dose dependent on patient response. Start at 2mIU/min, increasing every 30 minutes by 2mIU/min, to max 24mIU/min.

SUMMARY:
The purpose of this study is to examine the feasibility of using intracervical balloon catheters for cervical ripening as part of labour induction in healthy, GBS-negative women with prelabour rupture of membranes at term.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing two methods of induction of labour for pregnant, GBS-negative women presenting with prelabour rupture of membranes at term.

The intervention consists of the insertion of a double-balloon intracervical catheter at the time of induction, followed immediately by oxytocin infusion. The control consists of standard therapy: oxytocin induction. Our primary outcome is feasibility, and our secondary outcomes are length of first and second stages of labour, rate of vaginal delivery, intrapartum fever, chorioamnionitis, NICU admission, suspected or proven neonatal sepsis, or serious neonatal complication.

ELIGIBILITY:
Inclusion Criteria:

* Singleton Pregnancy
* 37.0 and 41.0 gestational age
* Confirmed Rupture of Membranes
* Group B Streptococcus Negative
* Cephalic Presentation
* Absence of contractions for at least 60 minutes following rupture
* Absence of contractions at time of enrolment

Exclusion Criteria:

* Contraindication to Vaginal Delivery
* Previous Uterine Surgery, including Caesarean Section
* Previous Cerclage, Cone Biopsy, LEEP, or Cervical Surgery
* Documented history of cervical incompetence
* High Grade intraepithelial lesion, adenocarcinoma in situ, or invasive cervical cancer.
* Immunosuppressed State
* Active Vaginal Infection

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Feasibility | 48 hours

SECONDARY OUTCOMES:
Intrapartum Fever | 48 Hours
Duration of Labour | 48 hours
NICU Admission | 0-7 days postpartum
Chorioamnionitis | 48 Hours
Patient Satisfaction | 0-6 weeks Postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Costescu, MD, BSc, Principal Investigator — McMaster University, Department of Obstetrics and Gynaecology; Amie Cullimore, MD BSc BEd, Principal Investigator — McMaster University, Department of Obstetrics and Gynaecology
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Costescu DJ, Cullimore AJ. Lessons learned from a resident-led clinical trial in obstetrics. Clin Trials. 2013 Aug;10(4):612-6. doi: 10.1177/1740774513492045. Epub 2013 Jun 13. PMID 23766376